CLINICAL TRIAL: NCT06347237
Title: PsA Digital Phenotyping and Inflammation Drivers Study
Acronym: PDPID
Status: Not yet recruiting | Type: Observational
Sponsor: Jolanda Luime (Other)
Collaborators: University of Oxford - Nuffield Department of Orthopaedics, Rheumatology and Musculoskeletal Sciences (Unknown); Aristotle University Of Thessaloniki (Other); Portuguese Society of Rheumatology - The Rheumatic Diseases Portuguese Registry (Reuma.pt) (Unknown)
Responsible Party: Sponsor-Investigator, Jolanda Luime, Principle investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL84429.078.23
Record Dates: First submitted 2024-02-14; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Psoriatic Arthritis; Flare Up, Symptom; Psoriatic Arthritis Aggravated
Keywords: psoriatic arthritis; inflammation; digital biomarker; flare
MeSH Terms: conditions — Arthritis, Psoriatic; Symptom Flare Up; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to develop and internally validate a machine learning model for detecting flare using a digital biomarker and a machine learning model for predicting flare, in patients with psoriatic arthritis. The main questions it aims to answer are:

* In patients with psoriatic arthritis, is a digital biomarker capable of detecting a flare as compared to clinical defined flare by the rheumatologist?
* In patients with psoriatic arthritis, what factors trigger a psoriatic arthritis flare ?

Participants will be requested to:

* Install app on their phone
* Use a smartwatch
* Complete questionnaires
* Collect biological material

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PsA
* Age 18 years or older and competent
* Using a smartphone
* Agree to use smartwatch
* Good command of the local language

Exclusion Criteria:

* Less than 18 years of age
* Incapacitated

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with psoriatic arthritis
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Absence of flare in patients | 12 months (follow-up every 3 months)
  Flare in psoriatic arthritis evaluated as:
  Patients
  * 'At this time, is your psoriatic arthritis in remission, if this means: you feel your disease is as good as gone?' yes/ no (for remission)
  * 'At this time, are you in low disease activity, if this means: your disease is in low activity but it's not as good as gone?' yes/ no (for low disease activity)
  Patient Acceptable Symptom State
  - 'If you were to remain for the next few months as you were during the last 48 hours, would this be acceptable or unacceptable for you?' yes/ no
  Doctors
  * 'At this time, is the psoriatic arthritis in remission, if this means: the absence of clinical and laboratory evidence of significant inflammatory disease activity?' yes/ no (for remission)
  * 'At this time, is the psoriatic arthritis in low or minimal disease activity?' yes/ no (for low disease activity)

SECONDARY OUTCOMES:
Minimal disease Activity (MDA) | 12 months (follow-up every 3 months)
  MDA as defined by patient meeting 5 out of 7 of the following criteria: (i) tender joint count ≤1; (ii) swollen joint count ≤1; (iii) Psoriasis Area and Severity Index ≤ 1 or body surface area ≤3%; (iv) tender entheseal points ≤ 1 (v) patient pain visual analogue scale VAS ≤15; (vi) patient global activity VAS ≤20; (vii) Health Assessment Questionnaire (HAQ) ≤0.5
Psoriatic Arthritis Disease Activity Score (PASDAS) | 12 months (follow-up every 3 months)
  PASDAS calculated as a composite score using the following criteria: physician global VAS, patient global VAS, SF36 physical (PCS), swollen joint count, tender joint count, Leeds Enthesitis Index, tender dactylitis count, and CRP. Higher scores indicate higher disease activity.
Disease Activity Psoriatic Arthritis (DAPSA) | 12 months (follow-up every 3 months)
  DAPSA calculated as a summation score of the following: tender and swollen joints, patient global assessment VAS, patient pain VAS and C-reactive protein. Higher scores indicate higher disease activity.
Psoriatic Arthritis Impact of Disease (PsAID) | 12 months (follow-up every 3 months)
  PsAID:10-point Likert scale questions on 12 items (pain, fatigue, skin, work/leisure activities, functional capacity, discomfort, sleep, coping, anxiety, embarrassment, social life, depression). Higher score indicates higher impact of disease.
Morning stiffness | 12 months (follow-up every 3 months)
  Morning stiffness on a 10-point Likert scale. Higher scores indicate higher morning stiffness.

OTHER OUTCOMES:
Keystroke dynamics | Continuous throughout 12 months
  Keypad time-related data and metadata collected unobtrusively from smartphone of patient
Screen time | Continuous throughout 12 months
  Screen time (hours) metrics collected unobtrusively from smartphone of patient
Accelerometer data | Continuous throughout 12 months
  Accelerometer data collected unobtrusively from smartphone of patient and smartwatch to measure physical activity. Patients will wear the smartwatch daily
Gyroscope sensor data | Continuous throughout 12 months
  Gyroscope sensor data for orientation collected unobtrusively from smartphone of patient
Steps count | Continuous throughout 12 months
  Count of steps collected unobtrusively from the smartwatch of patient to measure physical activity. Patients will wear the smartwatch daily
Physical activity intensity and categories | Continuous throughout 12 months
  Physical activity intensity and physical activity categories collected unobtrusively from the smartwatch of patient to measure physical activity. Intensity and categories are features provided by the smartwatch. Patients will wear the smartwatch daily
Motion | Continuous throughout 12 months
  Motion intensity collected unobtrusively smartwatch of patient to measure physical activity. This is a feature provided by the smartwatch. Patients will wear the smartwatch daily
Distance | Continuous throughout 12 months
  Distance (km) collected unobtrusively from smartwatch of patient to measure physical activity. Patients will wear the smartwatch daily
Pulse Ox | Continuous throughout 12 months
  Pulse Ox collected unobtrusively from smartwatch of patient to measure physical activity. Patients will wear the smartwatch daily
Respiration | Continuous throughout 12 months
  Respiration rate collected unobtrusively from smartwatch of patient to measure physical activity. Patients will wear the smartwatch daily
Body battery | Continuous throughout 12 months
  Body battery collected unobtrusively from smartwatch of patient to measure stress on a scale. This is a feature provided by the smartwatch. Patients will wear the smartwatch daily
Stress (digital) | Continuous throughout 12 months
  Stress levels collected unobtrusively from smartwatch of patient to measure stress on a scale. This is a feature provided by the smartwatch. Patients will wear the smartwatch daily
Heart rate | Continuous throughout 12 months
  Heart rate collected unobtrusively from smartwatch of patient to measure stress
Beat-to-beat intervals | Continuous throughout 12 months
  Beat-to-beat intervals collected unobtrusively from smartwatch of patient to measure stress
Sleeping time | Continuous throughout 12 months
  Sleeping time (hours) collected unobtrusively from smartwatch of patient
Sleeping type | Continuous throughout 12 months
  Sleeping type (%) collected unobtrusively from smartwatch of patient
Hand and feet photos | 12 months (follow-up every 6 weeks and in case of flare)
  Images of hands and feet of the patient captured by the smartphone camera of the patient, to produce a feature vector relative to the condition of nails and joints of hands and toes resulting in an imaging digital biomarker
Hand and body movements videos | 12 months (follow-up every 6 weeks and in case of flare)
  Videos of pre-specified movements of hand and body recorded by the smartphone camera of the patient, to produce a set of time series with landmark coordinates (obtained from the videos) resulting in an imaging digital biomarker
Medical history | 12 months (follow-up every 3 months)
  * Age (years)
  * Sex
  * Years of disease (years)
  * Medication over the year of the study
  * Comorbidity
  * Care activities
  * Job title, shift work
  * Frequent flying (days)
Joint count | 12 months (follow-up every 3 months)
  66/68 joint count for swelling and tenderness. Higher count indicates higher swollen/tender joints.
Enthesitis | 12 months (follow-up every 3 months)
  6 tendon count for enthesitis using Leeds Enthesitis Index
Body surface area | 12 months (follow-up every 3 months)
  Body Surface Area for skin
Weight | Baseline
  Weight (kg) to calculate body mass index (BMI)
Height | Baseline
  Height (cm) to calculate BMI
Abdominal circumference | Baseline
  Abdominal circumference (cm)
ClASsification criteria for Psoriatic ARthritis (CASPAR) score | Baseline
  CASPAR score calculation for the classification of PsA using points from the following criteria: (i) evidence of current psoriasis, or personal or family history of psoriasis, (ii) dactylitis, (iii) juxtaarticular new bone formation, (iv) nail dystrophy, and (v) negative for rheumatoid factor.
Demographics | 12 months (follow-up every 3 months)
  Questionnaire to assess demographics
VAS Pain | 12 months (follow-up every 3 months)
  VAS for pain assessment. Higher score indicate higher pain levels.
HAQ questionnaire | 12 months (follow-up every 3 months)
  HAQ questionnaire to measure physical function
VAS patient global | 12 months (follow-up every 3 months)
  VAS for patient global assessment
PSAID questionnaire | 12 months (follow-up every 3 months)
  PSAID questionnaire to measure impact of disease. Higher score indicates higher impact of disease.
SF-36 questionnaire | 12 months (follow-up every 3 months)
  SF-36 questionnaire for general health assessment
EQ5d questionnaire | 12 months (follow-up every 3 months)
  EQ5d questionnaire for general health assessment
Work Productivity and Activity Impairment (WPAI) questionnaire | 12 months (follow-up every 3 months)
  WPAI questionnaire for work impairment
Health care questionnaire | 12 months (follow-up every 3 months)
  Health care questionnaire for health care usage
Patient Health Questionnaire (PHQ9) questionnaire | 12 months (follow-up every 3 months)
  (PHQ9) questionnaire for depression assessment
Perceived Stress Scale (PSS) | 12 months (follow-up every 3 months)
  PSS questionnaire for stress
Global Rating of Change (GRoC) Scale | 12 months (follow-up every 3 months)
  GRoC scale to evaluate change in disease activity.
Life events questionnaire | 12 months (Baseline and month 12)
  Life events questionnaire for life events
Digital literacy questionnaire | Baseline
  Digital literacy questionnaire for technology readiness
Inflammatory blood marker | 12 months (follow-up every 3 months)
  Blood C-reactive protein levels (ml/L)
Genetic variants | Baseline
  Salivary DNA analysis
Gut microbiome | 12 months (Baseline, in case of flare, and months 6 and 12 in subgroup of patients)
  Stool analysis to extract bacterial DNA using 16S sequencing
Stress (cortisol levels) | 12 months (follow-up every 3 months)
  Hair cortisol analysis to measure stress

REFERENCES:
- See also: iPROLEPSIS project website — https://www.iprolepsis.eu/